CLINICAL TRIAL: NCT03863964
Title: Tranexamic Acid Administered After Delivery: Maternal Pharmacokinetics, Pharmacodynamics, and Coagulation Status
Brief Title: Tranexamic Acid Pharmacokinetics During Postpartum Hemorrhage
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michaela Kristina Farber, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P003122
Record Dates: First submitted 2018-12-11; First posted 2019-03-05 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Postpartum Hemorrhage
Keywords: tranexamic acid; pharmacodynamics; pharmacokinetics; pregnancy; thromboelastometry
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: This is a pilot study to determine the pharmacokinetics/pharmacodynamics of tranexamic acid administered after delivery to patients at high risk for postpartum hemorrhage, and coinciding coagulation testing using ROTEM®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (13):
- plasma TXA and ROTEM test at 3 minutes (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 7 minutes (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 15 minutes (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 30 minutes (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 1 hour (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 1.5 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 2 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 2.5 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 3 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 3.5 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 4 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 4.5 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test
- plasma TXA and ROTEM test at 5 hours (Active Comparator): Blood test
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — 13 blood samples will be drawn: at 3 min, 7 min, 15 min, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, and 5h post-treatment with TXA. Blood samples will be processed for ROTEM® analysis and for plasma concentration of TXA. TXA plasma concentrations will be modeled with a non-linear mixed-effects strategy using Monolix 4.1 and NONMEM(®) 7.2.

SUMMARY:
Postpartum hemorrhage (PPH) accounts for 20-25 percent of maternal deaths worldwide. Tranexamic Acid (TXA) is an antifibrinolytic agent that has been shown to reduce the estimated blood loss after delivery and is recommended by the World Health Organization for PPH treatment. However, dosing in studies ranges from 0.5g to 4g and the optimal dose of TXA in the pregnant population has not been established. Further, the effect of TXA on global coagulation assessed by rotational thromboelastometry (ROTEM®) has not been elucidated.

The primary aim of this study is to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of TXA administered after delivery in patients at risk for PPH.

DETAILED DESCRIPTION:
PPH occurs in approximately 1-5% of deliveries in the United States and accounts for 20-25% of maternal deaths worldwide. PPH is difficult to predict, but classically, risk factors for PPH- uterine atony, abruption, retained tissue, lacerations, infection, obesity, preeclampsia, magnesium administration, and prolonged labor- impede uterine contraction, vasoconstriction, and clotting. In addition, 40% of PPH occurs in the absence of known risk factors.

Early recognition of significant bleeding, pharmacologic therapy, and correction of coagulopathy are critical measures to minimize morbidity and mortality from PPH. TXA is an antifibrinolytic agent that competitively inhibits plasminogen, preventing activation of plasmin and lysis of fibrin. TXA is used in many surgical arenas including cardiac, orthopedic, pediatric, urologic, and gynecologic surgery and has been shown to be a useful adjunct to uterotonics to reduce blood loss after vaginal or cesarean delivery without maternal adverse effects.

The efficacy and side-effect profile of TXA is dose-dependent, but the optimal dose based on the pharmacokinetics (PK) and pharmacodynamics (PD) of TXA have yet to be determined in the obstetric population. Doses given after delivery have ranged from 0.5 to 4g bolus with or without a subsequent infusion. The World Maternal Antifibrinolytic (WOMAN) trial was a multi-country placebo-controlled randomized trial of 20,060 women in which placebo or TXA 1g IV over 10 minutes was administered at the onset of PPH, with a second dose (placebo or 1g TXA) if bleeding was ongoing at 30 minutes. Women who received TXA had a lower number of laparotomies and no increase in thromboembolic events including pulmonary embolus, myocardial infarction, and cerebral vascular accident. Women who received TXA less than 1 hour or greater than 3 hours after birth had similar risks of hysterectomy or death, but women who received TXA 1 to 3 hours after birth had a lower risk of hysterectomy or death from bleeding (World Health Organization; WHO). The 1g dose in the WOMAN trial was modeled after the Clinical Randomization of an Antifibrinolytic in Significant Haemorrhage (CRASH-2) trial, in which TXA was administered to trauma patients with hemorrhage. A French multicenter trial randomized 152 women to receive either 4g of TXA administered over 1 hour followed by a maintenance dose of 1g/hour for 6 hours, or standard care without TXA. Patients who received 10g TXA had reduced EBL, enhanced response to uterotonic agents, less change in hemoglobin values, lower number of blood products transfused, and a trend toward a lower rate of invasive surgical procedures. In the pediatric population, a wide range of TXA doses from 10mg/kg to 100mg/kg have been reported, with higher dose correlating with a reduction in blood loss, but also an increase in neurologic or thromboembolic complications.

Side effects from TXA are rare and include allergic reaction, dizziness, low blood pressure, nausea/vomiting, diarrhea, muscle spasm, and vision change. Serious potential complications associated with higher doses of TXA such as those used during cardiac surgery include thrombosis and seizures. However, TXA administered at lower doses for bleeding (1g to 2g IV, or a 10mg/kg bolus) is not associated with an increased rate of thrombosis or seizure activity. Given the potential seizure risk, the use of TXA in patients with a seizure disorder or in conditions that lower the seizure threshold such as preeclampsia may be relatively contraindicated, as TXA also lowers the seizure threshold through competitive antagonism of the inhibitory neurotransmitter glycine.

ROTEM® is a whole blood point-of-care assay of coagulation. There are anticipated hypercoagulable changes in the blood at term gestation and unpredictable changes in coagulation during PPH, making ROTEM® a potentially useful tool. The effect of TXA on maternal coagulation profile after delivery assessed by ROTEM® is unknown. The use of ROTEM® during TXA therapy in correlation with plasma TXA levels may help characterize the optimal dose for its impact on the coagulation profile. Further, it may help explain why in the WOMAN trial the most effective dosing time was between one and three hours after onset of PPH.

This study proposes to evaluate the PD and PK of TXA administered after delivery, in conjunction with its impact on coagulation measured by ROTEM®. The 2017 WHO Executive Guideline Steering Group on maternal and perinatal health recommends early use of TXA, within 3 hours of birth, for women with PPH (strong recommendation, moderate quality of evidence). TXA administration is therefore increasingly common during PPH. It is meaningful to explore the optimal dose of TXA that balances efficacy and safety: optimizing maternal TXA exposure (serum level) while minimizing the risk of thrombosis (increased hypercoagulable changes on ROTEM®).

ELIGIBILITY:
Inclusion Criteria:Age 18 and 50 years, gestational age > to 23 weeks at the time of admission for labor and delivery, and normal serum creatinine (< 0.9). Patients having either vaginal or cesarean delivery are eligible. Patients must have (1) major or (2 or more) minor risk factors for PPH as described here:

Major (1) or more:

* Suspected abnormal placentation
* Placenta previa
* Known coagulopathy
* Active concern for bleeding per care team

Minor (2) or more:

* 2 prior cesarean deliveries
* 3 prior deliveries
* Prior history of PPH
* Chorioamnionitis
* Polyhydramnios
* Macrosomia
* Obesity
* Suspected placental abruption

Exclusion Criteria:

* Allergy to tranexamic acid, inherited thrombophilia, history/current/intrapartum venous thrombosis, seizure disorder, renal or liver dysfunction, preeclampsia, anticoagulation therapy, or category III fetal heart rate tracing.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
TXA plasma concentration at baseline | baseline (before delivery, before treatment with TXA)
  measured by ultra-performance liquid chromatography and mass spectometry
TXA plasma concentration 15 minutes after treatment | after TXA administration: 15 minutes
  measured by ultra-performance liquid chromatography and mass spectometry
TXA plasma concentration 30 minutes after treatment | after TXA administration: 30 minutes
  measured by ultra-performance liquid chromatography and mass spectometry
TXA plasma concentration 1 hour after treatment | after TXA administration: 1 hour
  measured by ultra-performance liquid chromatography and mass spectometry
TXA plasma concentration 1.5 hours after treatment | after TXA administration: 1.5 hours
  measured by ultra-performance liquid chromatography and mass spectometry
TXA plasma concentration 2 hours after treatment | after TXA administration: 2 hours
  measured by ultra-performance liquid chromatography and mass spectometry
TXA plasma concentration 2.5 hours after treatment | after TXA administration: 2.5 hours
  measured by ultra-performance liquid chromatography and mass spectometry

SECONDARY OUTCOMES:
Rotational Thromboelastometry (ROTEM®) coagulation test at baseline | baseline (before delivery, before treatment with TXA)
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays
Rotational Thromboelastometry (ROTEM®) coagulation test at 15 minutes | after TXA administration: 15 minutes
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays
Rotational Thromboelastometry (ROTEM®) coagulation test at 30 minutes | after TXA administration: 30 minutes
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays
Rotational Thromboelastometry (ROTEM®) coagulation test at 1 hour | after TXA administration: 1 hour
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays
Rotational Thromboelastometry (ROTEM®) coagulation test at 1.5 hours | after TXA administration: 1.5 hours
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays
Rotational Thromboelastometry (ROTEM®) coagulation test at 2 hours | after TXA administration: 2 hours
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays
Rotational Thromboelastometry (ROTEM®) coagulation test at 2.5 hours | after TXA administration: 2.5 hours
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays
Rotational Thromboelastometry (ROTEM®) coagulation test at 3 hours | after TXA administration: 3 hours
  maternal blood will be evaluated with ROTEM EXTEM and FIBTEM assays

CONTACTS AND LOCATIONS:
Overall Officials: Michaela K Farber, MD MS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States